CLINICAL TRIAL: NCT01439685
Title: Comparison of Biliary Stenting Alone vs. Stenting With Photodynamic Therapy During Endoscopic Retrograde Cholangiopancreatography (ERCP): A Retrospective and Prospective Analysis
Brief Title: Comparison of Biliary Stenting Alone vs. Stenting With Photodynamic Therapy (PDT) During ERCP
Acronym: PDT
Status: Withdrawn | Type: Observational
Why Stopped: A single cohort, alternative trial was started.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1106011779
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; PDT; Photodynamic Therapy; Bile Duct; Bile Duct Obstruction; Jaundice; Biliary Stent; ERCP; Obstructive Jaundice
MeSH Terms: conditions — Cholangiocarcinoma; Cholestasis; Jaundice; Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biliary Stent plus Photodynamic therapy: Biliary Stent plus Photodynamic therapy
- Biliary Stent group: Biliary Stent group

SUMMARY:
This study entails retrospective and prospective review of data from a database protocol. Data gathered will be then analyzed for a set amount of patients. In this study, the investigators will compare biliary stenting vs. biliary stenting plus photodynamic therapy (PDT) and assess if PDT can improve quality of life and prolong survival.

DETAILED DESCRIPTION:
Successful palliation of biliary obstruction is the main goal for reducing morbidity and mortality in patients with biliary disease and biliary obstruction related to cholangiocarcinoma. Surgical biliary bypass is unfortunately complicated by a 30-day postoperative mortality rate of between 7 and 24%. Moreover, because of recovery time the quality of life following surgery is only improved in a minority. At present endoscopic insertion of a plastic or metal stent is the method of choice to relieve obstructive jaundice without the high morbidity and mortality associated with surgery. But this relief is unfortunately temporary since stents tend to become obstructed and the fact that effective biliary drainage in the proximal lesion is challenging. Photodynamic Therapy (PDT) is a new therapeutic approach that specifically targets neoplastic cells. This therapy involves the intravenous administration of a photosensitizing agent followed by activation of the agent by illumination with non-thermal light of a specific wavelength, resulting in cell death from direct cytotoxicity and ischemic necrosis. Cytotoxicity is directly proportional to tissue oxygenation.

A prospective, randomized and controlled trial study by Ortner et all confirmed the significant advantage of PDT with regard to relief of jaundice, quality of life, and survival. The improvement of survival in the randomized PDT group was so impressive that it was believed unethical to continue with randomization after the first 39 patients (20 and 19 in each group).Previously, the principal investigator conducted such a study (and also conducted Endoscopic Retrograde Cholangiopancreatography with PDT) at the University of Virginia, and would continue to conduct these procedures, as well as the study at WCMC.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone ERCP (Endoscopic Retrograde Cholangiopancreatography) and Biliary stenting with or without Photodynamic Therapy.
* Biliary disorder or obstruction due to Cholangiocarcinoma.
* Above 18 years of age.

Exclusion Criteria:

* Any patient who has not undergone ERCP and biliary stenting.
* Not diagnosed with Cholangiocarcinoma.
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from Cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of days patients survived post treatment | 2 years
  The group that receives PDT plus stenting will be compared to the group that received stenting only and their survival duration would be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Talreja JP, Kahaleh M. Photodynamic therapy for cholangiocarcinoma. Gut Liver. 2010 Sep;4 Suppl 1(Suppl 1):S62-6. doi: 10.5009/gnl.2010.4.S1.S62. Epub 2010 Sep 10. PMID 21103297
- [Result] Talreja JP, DeGaetani M, Sauer BG, Kahaleh M. Photodynamic therapy for unresectable cholangiocarcinoma: contribution of single operator cholangioscopy for targeted treatment. Photochem Photobiol Sci. 2011 Jul;10(7):1233-8. doi: 10.1039/c0pp00259c. Epub 2011 Apr 21. PMID 21512706